CLINICAL TRIAL: NCT07039461
Title: Evaluation of Effectiveness and Safety of Intense Pulsed Light Treatment for Chalazion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: identification of several protocol deviations that may affect the primary outcome accuracy
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUM-VBU-OPT-25-01
Record Dates: First submitted 2025-06-09; First posted 2025-06-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Chalazion
MeSH Terms: conditions — Chalazion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Study arm (Experimental): subjects in the study arm will receive active IPL treatment
  Interventions: Device: OptiLIGHT
- Control arm (Sham Comparator): subjects in the control arm will receive sham IPL treatment
  Interventions: Device: OptiLIGHT

INTERVENTIONS:
Device: OptiLIGHT — three IPL or sham treatment in 1 week interval followed by 1 follow-up 4 weeks after the last treatment

SUMMARY:
To study the effectiveness and safety of IPL treatment for Chalazion

DETAILED DESCRIPTION:
The study aims to evaluate the effectiveness and safety of IPL therapy for the treatment of chalazion. The effect of IPL on chalazion will be examined in a masked randomized controlled study. Subjects in the study arm will be treated with IPL, while subjects in the control arm will be treated with sham IPL. A significant difference in the outcomes of the two arms will provide support for a genuine contribution of the IPL treatment

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to read, understand, and sign an Informed Consent Form (ICF)
* 18 years of age or older
* Clinical diagnosis of acute chalazion, present for a maximum of 4 weeks
* Subject is willing to comply with all study procedures

Exclusion Criteria:

* Subjects who underwent IPL treatment less than 6 months prior to screening
* Concurrent eyelid infection, which to the opinion of the study investigator is not related to the chalazion
* Chalazion with atypical features, which to the opinion of the study investigator is inadequate for a study
* Chronic Chalazion
* Recurring Chalazion
* Floppy eyelid syndrome
* Demodex blepharitis patients taking Lotilaner ophthalmic solution within 30 days prior to screening
* Ocular surgery within 3 months prior to screening
* Current diagnosis of malignant tumors in the affected eyelid, including: sebaceous carcinoma and basal cell carcinoma
* Laser Assisted In Situ Keratomileusis (LASIK)/Small Incision Lenticule Extraction (SMILE) surgery, within 1 year prior to screening
* Radial Keratotomy (RK) surgery
* Recent ocular trauma, within 3 months prior to screening
* Pre-cancerous lesions or skin cancer in the planned treatment area
* Severe active allergies, or other severe uncontrolled eye disorders affecting the ocular surface
* Uncontrolled infections or uncontrolled immunosuppressive diseases
* Best corrected visual acuity worse than 20/200 in either eye
* Ocular surface abnormality that may compromise corneal integrity in either eye (e.g., prior chemical burn, Epithelial Basement Membrane Dystrophy - EBMD)
* Within 3 months prior to screening, use of photosensitive medication and/or herbs that may cause sensitivity to 560-1200 nm light exposure, including: Isotretinoin, Tetracycline, Doxycycline, and St. John's Wort
* Active sun burn in the treatment area
* Anterior chamber inflammation
* Corneal edema
* Any condition revealed whereby the investigator deems the subject inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2025-09-12 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2025-12-24 (Actual)

PRIMARY OUTCOMES:
The percentage of resolved chalazion 4 weeks after the last treatment in the study group and the control group | 4 weeks after the last treatment
  the proportion of subjects with reduction of at lease 80% in lesion size at the follow up visit

SECONDARY OUTCOMES:
Percentage change from baseline in lesion size in both groups | 4 weeks after the last treatment
  measuring the lesion size using a millimeter ruler
Time to resolution which is defined as a reduction of at least 80% in lesion size in both groups | 4 weeks after last treatment
  measuring the time that takes for a reduction of at least 80% in lesion size

OTHER OUTCOMES:
modified Meibomian Gland Score | 4 weeks after the last treatment
  15 Meibomian glands along the lower lid (5 nasal + 5 central + 5 temporal) will be gently expressed with the dedicated expression forceps. Each gland will be scored 0 to 3, as follows: 0 = clear liquid meibum; 1 = cloudy liquid meibum; 2 = inspissated meibum; 3 = blocked). The modified Meibomian Gland score will be evaluated as the sum of scores for these 15 glands. Hence, the minimal value is 0 (all 15 glands express a clear liquid meibum), and the maximal value is 45 (all 15 glands are blocked). A decrease in the modified Meibomian Gland Score means that the functionality of Meibomian glands improved, and that the condition of the patient improved.
Teat Breakup time | 4 weeks after the last treatment
  Time between full blink and first appearance of a break in a fluorescein-stained eye
BCVA | 4 weeks after the last treatment
  Best-corrected visual acuity, using an ETDRS chart (20/20, 20/25, 20/32,20/40,20/50,20/63, 20/80, 20/100, 20/200, 20/400, where 20/20 is considered perfect vision and 20/400 is considered legal blindness)
Adverse events | Throughout the study and up to 4 weeks after the last treatment
  Incidence and type of adverse events
Pain/Discomfort | day 0, day 7, day 14
  Pain/discomfort will be self-reported with a visual analog scale (0 to 10), with 0 representing no pain/discomfort and 10 representing intolerable pain/discomfort.
IOP | 4 weeks after the last treatment
  intra ocular pressure using tonometer
Biomicroscopy | 4 weeks after the last treatment
  Eyelid appearance will be assessed with biomicroscopy at the slit lamp
satisfaction level | 4 weeks after the last treatment
  subject will fill out a satisfaction questionnaire (very satisfied/satisfied/neutral/disappointed/very disappointed).

CONTACTS AND LOCATIONS:
Overall Officials: James Chelnis, MD, Principal Investigator — Manhattan Face and Eye; Laura Periman, MD, Principal Investigator — Periman Eye Institute
Locations (2):
- United States (2):
  - Manhattan Face and Eye clinic, New York, New York
  - Periman Eye Institute, Seattle, Washington